CLINICAL TRIAL: NCT05681390
Title: A Prospective, One-arm, Phase II Clinical Study of Tislelizumab Combined With Anlotinib and Investigator-selected Chemotherapy for Second-line Treatment of Advanced or Metastatic Pancreatic Cancer: a
Brief Title: Tislelizumab With Anlotinib and Chemotherapy for Second-line Treatment of Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSL-010X1
Record Dates: First submitted 2022-12-09; First posted 2023-01-12 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Neoplasms
Keywords: Advanced; second-line treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab Combined With Anlotinib and Chemotherapy (Experimental): Tislelizumab iv drip, every 3 weeks; Anlotinib, oral，once a day; chemotherapy will be choiced by investigator according guildline.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg iv drip, d1, Q3W;Anlotinib tablet : 10mg, PO, QD; Chemotherapy: selected by investigator following CSCO or NCCN pancreatic adenocarcinoma guideline; Tislelizumab and Anlotinib continue unless disease progression or intolerance to toxicity, chemotherapy continue upto 8 cycles unless disease progression or intolerance to toxicity
  Other Names: Beigene

SUMMARY:
This is a prospective, one-arm, phase II clinical study of Tislelizumab Combined With Anlotinib and Chemotherapy for Second-line Treatment of Advanced or Metastatic Pancreatic Cancer

DETAILED DESCRIPTION:
This is a single-arm, open-label, clinical trial of tislelizumab in combination with anlotinib and investigator-selected chemotherapy for second-line treatment of patients with advanced or metastatic pancreatic cancer. Patients with histopathologically or cytologically confirmed unresectable, recurrent or metastatic pancreatic cancer are planned to be recruited. Systemic medical antineoplastic therapy previously treated with first-line chemotherapy, meeting the inclusion and exclusion criteria of this study, and giving tislelizumab and anlotinib in combination with investigator 's choice of second-line chemotherapy regimen

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic pancreatic adenocarcinoma diagnosed by pathology;
* Previously received a standard first-line chemotherapy regimen of pancreatic cancer
* Age ≥ 18 and≤ 75 years old;
* Expected survival ≥ 3 months;
* ECOG score 0-1;
* Child-Pugh score < 8;
* There is at least one measurable tumor lesion: the long diameter is ≥10 mm, and the short diameter of lymph nodes is ≥15 mm;
* The results of liver and kidney function and blood routine examination within 1 week before enrollment meet the following conditions:

Neutrophils (ANC) ≥ 1.5×109/L, platelets (PLT) ≥ 80×109/L, hemoglobin (HGB) ≥ 80g/L; Serum creatinine (Cr) ≤ 1.5 × upper limit of normal value; total bilirubin (TBIL) ≤ 2.5 × upper limit of normal value, Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤2.5× upper limit of normal value;

- The patient voluntarily participated in this study and signed the informed consent form.

Exclusion Criteria:

* Received other immunotherapy previously(including immune checkpoint inhibitor PD-1/PDL1 and other immune checkpoint inhibitors) and/or anti-angiogenic drugs (including anti-VEGFR monoclonal antibody and anti-angiogenic small molecule kinase inhibitors) ; Known to be severely allergic to the drugs used in the study of tislelizumab and anlotinib;
* Patients with obstructive jaundice who cannot reach TBIL ≤ 2.5 times the upper limit of normal value after surgical intervention;
* Patients with biliary obstruction that may occur or worsen within 4 to 6 weeks;
* Obvious blood coagulation disorder, active bleeding and bleeding tendency;
* There is a history of other malignant tumors within 5 years (adequately treated skin basal cell carcinoma, cervical in situ);
* Interstitial pneumonia or pulmonary fibrosis;
* Uncontrollable pleural effusion or ascites;
* Severe uncontrolled medical diseases, acute infections, recent history of myocardial infarction (within 3 months);
* During pregnancy or breastfeeding, and those who refuse to take appropriate contraceptive measures during the test;
* Patients judged by the investigator to be inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
MedianProgression free survival(mPFS) | from enrollment to disease progression or death from any cause, up to 24 months
  assessment by RECIST v1.1,at end of per 2 treatment cycles(each cycle is 21 days)

SECONDARY OUTCOMES:
objective response rate(ORR) | from enrollment to disease progression or death from any cause,up to 24 months
  assessment by RECIST v1.1,at end of per 2 treatment cycles(each cycle is 21 days)
Median Overall Survival | from enrollment to death from any cause,up to 24 months
  document and assessment on baseline, at end of 2 treatment cycles(each cycle is 21 days）
disease control rate(DCR) | up to 24 months
  document and assessment on baseline, at end of 2 treatment cycles(each cycle is 21 days）

CONTACTS AND LOCATIONS:
Overall Officials: EnXiao Li, Doctor, Principal Investigator — First hospital of Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No